CLINICAL TRIAL: NCT04644861
Title: Evaluation of the Feasibility of a Physical Activity Program Adapted for Primary Care, for People Aged 70 and Over Who Have At Least One Long-term Illness
Brief Title: Adapted Physical Activity Centre (in The) CITY for Elders Aged 70 and Over with At Least One Long Term Illness
Acronym: CAPACITY70
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/19/0057; 2020-A01164-35 (Other: IDRCB)
Record Dates: First submitted 2020-11-03; First posted 2020-11-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Chronic Disease
Keywords: Chronic Disease; adapted physical activity; primary care; Motor Activity; Elders
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elders aged 70 (Other): Program of adapted physical activity
  Interventions: Other: Program of adapted physical activity

INTERVENTIONS:
Other: Program of adapted physical activity — 3 workouts of one hour every week during 4 months. Program will be conducted by adapted physical activity teachers and sports doctor.

SUMMARY:
Elders aged 70 and over, living in Toulouse, with a chronic disease identified by the French social insurance as an Affection Longue Durée will be eligible to a 4 months physical activity program in a primary health center. This program will be proposed by their general practitioner. The aim of the study is to establish the feasibility of such program conduced exclusively in primary care.

DETAILED DESCRIPTION:
The number of elders aged 70 and over and suffering of a chronic disease are increasing in our country. These patients are at risk of sarcopenia which can lead to an increasing risk of falls and hospitalization, loss of autonomy, and morbi-mortality. Twelve weeks adapted physical activity program can manage sarcopenia in elders. One of the difficulties to propose such a program to elders patients is the difficulty to reach the program center due to mobility deficiency. Our hypothesis is that proposing an adapted physical activity in a primary health care center, in the city of the patient, could help the participation.

Eligible patients addressed by their general practitioner will perform 4 months adapted physical activity program in the CAPA-CITY center (MSPU La Providence).

The inclusion will be realized by the sports doctor of CAPA-CITY. At M2, sport doctor and adapted physical activity teacher will meet the patient to readapt the program taking in count his particularity and wishes.

At M4 M6 and M12, an independent global evaluation will be realized by training nurse and clinical research associate.

ELIGIBILITY:
Inclusion Criteria:

* Elders aged 70 and over, with a chronic disease recognize as an Long Term Affection by the French social insurance.
* Living at home in Toulouse
* With a general practitioner working in Toulouse and agreed to participate to the CAPA-CITY70 program research

Exclusion Criteria:

* Elders living in nursing home
* Elders dependent for daily activity (score < 5.5 Autonomy scale of Katz)
* Elders with dementia according to DSM V criteria
* Elders participating in another research project
* Contraindication for physical activity

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
feasibility of the adapted physical activity program (ratio 1) | Month 0
  total number of patients included in the study
feasibility of the adapted physical activity program (ratio 2) | Month 4
  number of patients who complete the program of adapted physical activity in totality

SECONDARY OUTCOMES:
feasibility complementary criteria Month 0 | Month 0
  number of patients who start the program of adapted physical activity
feasibility complementary criteria Month 4 | Month 4
  reasons to not complete the program of adapted physical activity
organization feasibility | Month 4
  number of canceled sessions
program adhesion (sessions realised) | Month 4
  numbers of realised session
patient's quality of life measured by Whoqol-bref (World Health Organization Quality Of Life - Bref) | Month 0
  patient's quality of life measured by Whoqol-bref. Score from 0 to 100, higher score mean better outcome
patient's quality of life measured by Whoqol-bref (World Health Organization Quality Of Life - Bref) | Month 4
  patient's quality of life measured by Whoqol-bref. Score from 0 to 100, higher score mean better outcome
patient's quality of life measured by Whoqol-bref (World Health Organization Quality Of Life - Bref) | Month 12
  patient's quality of life measured by Whoqol-bref. Score from 0 to 100, higher score mean better outcome
patient's physical activity measured by GPAQ Global Physical Activity Questionnaire | Month 0
  Global Physical Activity Questionnaire (GPAQ). Score from 0 to 3000. higher score mean better outcome
patient's physical activity measured by GPAQ Global Physical Activity Questionnaire | Month 6
  Global Physical Activity Questionnaire (GPAQ), Score from 0 to 3000, higher score mean better outcome
patient's physical activity measured by GPAQ Global Physical Activity Questionnaire | Month 12
  Global Physical Activity Questionnaire (GPAQ), Score from 0 to 3000, higher score mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Emile ESCOURROU, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de TOULOUSE, Toulouse, France

IPD SHARING:
Plan to Share IPD: No